CLINICAL TRIAL: NCT05075239
Title: Incidence Of Morbidity And Mortality After Isolated Traumatic Brain Injury In Adult Neuro-intensive Care Unit In Minia University Hospital
Brief Title: Morbidity and Mortality in Solo Adult Traumatic Brain Injury Patients in Minia University Hospital
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Other Study IDs: 411-9/2021
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Statistical Analysis of Traumatic Brain Injury Victims
Keywords: neurotrauma; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tracking post-traumatic brain injury sequale

ELIGIBILITY:
Inclusion Criteria:

* Solo non penetrating neurotrauma victims

Exclusion Criteria:

* 1- Penetrating head trauma. 2- Polytrauma patients. 3- Coexist of Psychiatric disorders or history of neuronal disorders. 4- Refusal of patient relatives to participate in the assignment. 5- Pregnant females with TBI. 6- Patients who died during 24 hours from admission to ICU . 7- Patients more than 65 years of age .

  8- combined abdominal or orthopedic trauma.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: both sexes with individual neurotrauma
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
mortality and morbidity | 4 weeks
  number of deaths from neurotrauma

SECONDARY OUTCOMES:
prediction | one week
  to examine the predictors of outcome including age , gender , admission systolic blood pressure < 90 mmHg , GCS score ,APACHE II score ,lateralization of pupil , brain CT findings ,serum sodium &potassium ,mechanical ventilation and length of stay in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Maher Maher, Minya, Egypt, Egypt